CLINICAL TRIAL: NCT05001789
Title: Cognitive Functioning in Opioid Use Disorder: Examining the Impacts of Computerized Working Memory Training and Non-Fatal Opioid Overdose
Brief Title: Cognitive Functioning in Opioid Use Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NYSPI-wide Institutional Research Pause as of June 12, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Sandra D. Comer, Professor of Neurobiology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8185
Record Dates: First submitted 2021-07-09; First posted 2021-08-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use; Cognitive Change; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and research staff will be blinded to participant's training condition (active vs. sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Working memory training with task-difficulty increasing across sessions
  Interventions: Other: CogMed
- Sham (Active Comparator): Working memory training with task-difficulty remaining constant across sessions.
  Interventions: Other: CogMed

INTERVENTIONS:
Other: CogMed — 20 sessions of Cogmed working memory training

SUMMARY:
This outpatient study is designed to examine the potential relationship between non-fatal opioid overdose and cognitive functioning. This study will also examine the impact of computerized working memory training on relevant outcomes (cognition, psychosocial functioning, quality of life, drug use). The training component of the study lasts 1 month, with follow up visits and 1-month and 3-months post training.

DETAILED DESCRIPTION:
This outpatient study is designed to examine the potential relationship between non-fatal opioid overdose (i.e. overdose that does not result in death), cognitive functioning, and the impact of computerized working memory training on relevant outcomes (cognition, psychosocial functioning, quality of life). Participants (n=30) with a history of at least one prior opioid OD, who are enrolled in buprenorphine treatment, will be randomized to 20 sessions of an active (n=15) or sham (n=15) working memory training. Patients will complete measures of cognitive functioning during screening, post-training, and at 1-month and 3-month follow up. Participants will also complete the measures of decision making, psychosocial functioning and drug use at baseline, post-training, and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 criteria for moderate-severe Opioid Use Disorder (OUD) in the past 6 months
* Enrolled in a suboxone (buprenorphine/naloxone) program; willing to provide consent for research team to contact treatment provider
* History of at least 1 prior opioid overdose
* Recent history of illicit opioid use
* In good physical health
* Access to a smartphone, tablet, or computer

Exclusion Criteria:

* Evidence of a co-occurring, untreated psychiatric condition that would make participation risky or difficulty
* Lack of access to a home computer, smartphone, or tablet
* Unable to speak, read and/or communicate in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox Cognition Battery | Post-Training (1-month from baseline)
  A brief computerized test of key neuropsychological functions
NIH Toolbox Cognition Battery | 1-month Follow up
  A brief computerized test of key neuropsychological functions
NIH Toolbox Cognition Battery | 3-month Follow up
  A brief computerized test of key neuropsychological functions

SECONDARY OUTCOMES:
Psychosocial Functioning (Brief Inventory of Psychosocial Functioning B-IPF) | Post-training (1 month from baseline)
  B-IPF: scores range from 0 to 49 with higher scores indicating greater difficulties with psychosocial functioning
Psychosocial Functioning (Brief Inventory of Psychosocial Functioning B-IPF) | 1-month follow up
  B-IPF: scores range from 0 to 49 with higher scores indicating greater difficulties with psychosocial functioning
Psychosocial Functioning (Brief Inventory of Psychosocial Functioning B-IPF) | 3-month follow up
  B-IPF: scores range from 0 to 49 with higher scores indicating greater difficulties with psychosocial functioning
Illicit Substance Use: Timeline Follow Back (TLFB) | Post-training (1-month from baseline)
  TLFB: measures substance use in the past 1-week period
Illicit Substance Use: Timeline Follow Back (TLFB) | 1-month follow up
  TLFB: measures substance use in the past 1-week period
Illicit Substance Use: Timeline Follow Back (TLFB) | 3-month follow up
  TLFB: measures substance use in the past 1-week period
Quality of Life Scale (QOLS) | Post-training (1 month from baseline)
  QOLS: scores range from 16 to 112 with higher scores indicating greater quality of life
Quality of Life Scale (QOLS) | 1-month follow up
  QOLS: scores range from 16 to 112 with higher scores indicating greater quality of life
Quality of Life Scale (QOLS) | 3-month follow up
  QOLS: scores range from 16 to 112 with higher scores indicating greater quality of life
Impulsive decision making (Delay Discounting Task) | Post-training (1 month from baseline)
  Delay Discounting Task
Impulsive decision making (Delay Discounting Task) | 1-month follow up
  Delay Discounting Task
Impulsive decision making (Delay Discounting Task) | 3-month follow up
  Delay Discounting Task

CONTACTS AND LOCATIONS:
Locations (1):
- NY State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05001789/ICF_000.pdf